CLINICAL TRIAL: NCT01463982
Title: A Phase I Clinical Trial to Determine the Maximum Tolerated Dose and to Assess the Safety of OratecanTM in Combination With Capecitabine in Patients With Advanced Solid Cancer
Brief Title: Phase I of OratecanTM in Combination With Capecitabine in Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-OTE-103
Record Dates: First submitted 2011-10-31; First posted 2011-11-02 (Estimated); Results first posted 2015-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Solid Tumor; Advanced Cancer
Keywords: Advanced solid cancer
MeSH Terms: interventions — Capecitabine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oratecan and Capecitabine (Experimental): Oratecan(HM30181AK + Irinotecan HCl) and Capecitabine
  * Irinotecan HCl Tablet - Initial dose 10 mg/m2 (may be increased up to 20 mg/m2), Day1~Day5
  * HM30181AK Tablet - Fixed dose 15 mg, Day1~Day5
  * Capecitabine Tablet - Initial dose 800 mg/m2 (may be increased up to 1000 mg/m2), Day1~Day14
  Interventions: Drug: Oratecan and Capecitabine

INTERVENTIONS:
Drug: Oratecan and Capecitabine — Oratecan in combination with Capecitabine
  * Irinotecan HCl Tablet - Initial dose 10 mg/m2 (may be increased up to 20 mg/m2), Day1~Day5
  * HM30181AK Tablet - Fixed dose 15 mg, Day1~Day5
  * Capecitabine Tablet - Initial dose 800 mg/m2 (may be increased up to 1000 mg/m2), Day1~Day14
  Other Names: Oratecan(HM30181AK + Irinotecan HCl) and Capecitabine

SUMMARY:
The main objective of this study is to determine the maximum tolerated dose (MTD) of Oratecan in combination with capecitabine

DETAILED DESCRIPTION:
Besides the main objective, there are 4 other objectives as follows:

* To assess the safety of Oratecan in combination with capecitabine
* To evaluate anticancer activity of Oratecan in combination with capecitabine in patients with advanced solid malignancies
* To characterize the pharmacokinetics of Oratecan and its metabolites following oral administration of OratecanTM in combination with capecitabine

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced solid tumor
* Patients who have experienced progressive disease despite of conventional anticancer therapy. Patients who cannot expect effective treatment or prolonged survival with conventional anticancer therapy
* Previous chemotherapy, radiotherapy and surgical operation are allowed if they are discontinued for at least 4 weeks prior to D0 and all adverse events are resolved
* Aged ≥19
* Eastern Cooperative Oncology Group (ECOG) performance score of less than or equal to 2
* A life expectancy greater than 12 weeks
* Adequate bone marrow, renal and liver function.
* Subjects must provide written informed consent prior to performance of study specific procedures or assessments, and must be willing to comply with treatment and follow up assessments and procedures

Exclusion Criteria:

* Patients with hematopoietic malignancies,uncontrolled infection, CNS metastasis.
* Patients who have undergone hematopoietic stem cell transplantation (HSCT) or are candidates for planned HSCT
* Patients who have GI malabsorption or difficulty taking oral medication
* Patients who have psychiatric or congenital disorder Subjects who, in the investigator's opinion, cannot be treated per protocol due to functional impairments
* Pregnant or breast-feeding patients; Women of childbearing potential without adequate contraception (Men must use adequate contraception.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-12; Primary Completion 2012-04 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jina Jung, PhD, Study Director — Hanmi Pharmaceuticals.Co.,Ltd
Locations (1):
- Hanmi Pharmaceuticals, Co., Ltd, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Capecitabine 800mg/㎡ + Oratecan 10mg/㎡; Capecitabine 800mg/㎡ + Oratecan 15mg/㎡; Capecitabine 800mg/㎡ + Oratecan 20mg/㎡; Capecitabine 1000mg/㎡ + Oratecan 15mg/㎡: One cycle was composed of 3 weeks. Oratecan™ was administered once daily for 5 consecutive days, and Capecitabine Tablet was administered twice daily for 14 consecutive days, followed by washout period for 7 days.
Period: Overall Study
Arm/Group | Capecitabine 800mg/㎡ + Oratecan 10mg/㎡ | Capecitabine 800mg/㎡ + Oratecan 15mg/㎡ | Capecitabine 800mg/㎡ + Oratecan 20mg/㎡ | Capecitabine 1000mg/㎡ + Oratecan 15mg/㎡
Started | 3 | 8 | 4 | 6
Completed | 3 | 7 | 2 | 6
Not Completed | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Treatment delay over 5 week | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Capecitabine 800mg/㎡ + Oratecan 10mg/㎡ | Capecitabine 800mg/㎡ + Oratecan 15mg/㎡ | Capecitabine 800mg/㎡ + Oratecan 20mg/㎡ | Capecitabine 1000mg/㎡ + Oratecan 15mg/㎡ | Total
Number analyzed (Participants) | 3 | 8 | 4 | 6 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (6.5) | 59.5 (9.6) | 63.8 (11.1) | 61.8 (11.5) | 61.5 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 2 | 5
  Male | 3 | 6 | 3 | 4 | 16
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 3 | 8 | 4 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity Assessment and Maximum Tolerated Dose Determination
Description: If Dose Limiting Toxicity(DLT) was not observed in the third subject at a dose level from the first study drug dosing date (Day 1) to the end of Cycle 1(21 days), increase the dose to the next level and enroll subjects; enrollment up to Level 4 was allowed. (NCI-CTCAE version 3.0)
Time Frame: Cycle 1 (21 days)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Capecitabine 800mg/㎡ + Oratecan 10mg/㎡ | Capecitabine 800mg/㎡ + Oratecan 15mg/㎡ | Capecitabine 800mg/㎡ + Oratecan 20mg/㎡ | Capecitabine 1000mg/㎡ + Oratecan 15mg/㎡
Number analyzed (Participants) | 3 | 8 | 4 | 6
percentage of participants | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 36.9] | 50.0 [6.8 to 93.2] | 0.0 [0.0 to 45.9]

2. Secondary Outcome: Objective Response Rate (ORR), Response Rate (RR) and Disease Control Rate (DCR)
Description: by RECIST guideline Objective response rate = (Number of subjects with best overall response as confirmed CR or PR / Total number of subjects)*100.
  Response rate = (Number of subjects with best overall response as CR or PR / Total number of subjects)*100.
  Disease control rate = (Number of subjects with best overall response as confirmed CR or PR or SD / Total number of subjects)*100.
Time Frame: tumor response evaluation can continue to receive the study drug until PD confirmation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Capecitabine 800mg/㎡ + Oratecan 10mg/㎡ | Capecitabine 800mg/㎡ + Oratecan 15mg/㎡ | Capecitabine 800mg/㎡ + Oratecan 20mg/㎡ | Capecitabine 1000mg/㎡ + Oratecan 15mg/㎡
Number analyzed (Participants) | 3 | 7 | 2 | 6
percentage of participants
  Objective Response rate | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 84.2] | 33.3 [4.3 to 77.7]
  Response Rate | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 84.2] | 33.3 [4.3 to 77.7]
  Disease Control Rate | 66.7 [9.4 to 99.2] | 42.9 [9.9 to 81.6] | 100 [15.8 to 100.0] | 50.0 [11.8 to 88.2]

ADVERSE EVENTS:
Time Frame: From starting study medication to discontinuation of study medication
Description: The patient took study medication until meet withdrawal criteria.
Arm/Group | Capecitabine 800mg/㎡ + Oratecan 10mg/㎡ | Capecitabine 800mg/㎡ + Oratecan 15mg/㎡ | Capecitabine 800mg/㎡ + Oratecan 20mg/㎡ | Capecitabine 1000mg/㎡ + Oratecan 15mg/㎡
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/8 | 1/4 | 0/6
Other Adverse Events (participants affected / at risk) | 3/3 | 8/8 | 4/4 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine 800mg/㎡ + Oratecan 10mg/㎡ (N=3) | Capecitabine 800mg/㎡ + Oratecan 15mg/㎡ (N=8) | Capecitabine 800mg/㎡ + Oratecan 20mg/㎡ (N=4) | Capecitabine 1000mg/㎡ + Oratecan 15mg/㎡ (N=6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine 800mg/㎡ + Oratecan 10mg/㎡ (N=3) | Capecitabine 800mg/㎡ + Oratecan 15mg/㎡ (N=8) | Capecitabine 800mg/㎡ + Oratecan 20mg/㎡ (N=4) | Capecitabine 1000mg/㎡ + Oratecan 15mg/㎡ (N=6)
Diarrhoea (Gastrointestinal disorders) | 2 | 6 | 3 | 5
Nausea (Gastrointestinal disorders) | 2 | 6 | 4 | 3
Vomiting (Gastrointestinal disorders) | 2 | 4 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 4 | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 2 | 2 | 3
Pyrexia (General disorders) | 0 | 1 | 2 | 2
Oedema peripheral (General disorders) | 1 | 1 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 2
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator will complete the report on this study through discussion with Hanmi Pharmaceutical Co., Ltd. after the study is completed. If the report is to be published, prior agreement in writing should be made between the two parties.